CLINICAL TRIAL: NCT03722251
Title: Active Video-game Playing and a Glucose Preload on Food Intake Regulation in Children
Brief Title: Active Video-game Playing and Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB: 2012-120-1
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Appetitive Behavior
Keywords: appetite, food intake, active gaming
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: Repeated measures cross-over design.
Who Masked: Participant
Oversight: FDA-regulated Drug: No

ARMS (4):
- Glucose Beverage (Experimental): 50 g of glucose in solution
  Interventions: Behavioral: Glucose beverage, control beverage, glucose beverage and active video game playing, control beverage and active video game playing
- Control Beverage (Experimental): Sucralose in solution
  Interventions: Behavioral: Glucose beverage, control beverage, glucose beverage and active video game playing, control beverage and active video game playing
- Glucose beverage and active video game playing (Experimental): 50 g of glucose in solution and 30 min of active video game playing
  Interventions: Behavioral: Glucose beverage, control beverage, glucose beverage and active video game playing, control beverage and active video game playing
- Control Beverage and active video game playing (Experimental): Sucralose in solution and 30 min of active video game playing
  Interventions: Behavioral: Glucose beverage, control beverage, glucose beverage and active video game playing, control beverage and active video game playing

INTERVENTIONS:
Behavioral: Glucose beverage, control beverage, glucose beverage and active video game playing, control beverage and active video game playing

SUMMARY:
The purpose of this experiment is to investigate the effect of active video game playing for 30 minutes on food intake and subjective appetite. The investigators hypothesize that video game playing will affect food intake in children. Food intake will be measured at 30 minutes following a glucose (50g glucose in 250ml of water) or sweetened non-caloric (150mg Sucralose® in 250ml of water) beverage with or without active video game playing. Subjective appetite will be measured at 0, 15, 30 and 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

healthy boys with no emotional, behavioral or learning problems

Exclusion Criteria:

* Exclusion criteria are children with significant behavioral or emotional difficulties, those with dietary restrictions, or those taking medications.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2012-04-06 (Actual); Primary Completion 2015-05-25 (Actual); Study Completion 2015-05-25 (Actual)

PRIMARY OUTCOMES:
Food Intake (kcal) | 30 minutes after treatment
Subjective appetite (mm) | baseline and then 15, 30, and 60 minutes after preload consumption
  subjective appetite assessed by motivation-to-eat visual analogue scale. The scale range is between 0 and 100 mm. Higher scores represent higher appetite

SECONDARY OUTCOMES:
Subjective Mood (mm) | baseline and then 15, 30, and 60 minutes after preload consumption
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request.